CLINICAL TRIAL: NCT06159192
Title: Monitoring Effect Of Shock Wave On Microcirculation Changes In Type2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Head of the Department of Physiotherapy for Cardiovascular/ Rspiratory disorder and Geriatrics, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shock wave and neuropathy
Record Dates: First submitted 2023-11-20; First posted 2023-12-06 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Shock Wave and Nitric Oxide
Keywords: Shock Wave; Ntric oxide; Diabetes mellitus; Nerve conduction velocity
MeSH Terms: conditions — Diabetes Mellitus | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Monitor the effect of low intensity extracorporeal shock wave therapy on impaired nitric oxide synthase and microcirculation changes in type 2 diabetes mellitus with peripheral neuropathy
Who Masked: Participant
Masking Description: A group of 80 patients (male and female) diagnosed as type 2 diabetes mellitus, will be included in the study. Their age will be ranged from 40-60 years. Their weight ranged from 80 - 100 k.g. and their height ranged from 160 - 180 cm. Patients will divide into two groups: Study groups (A) 40 patients type 2 diabetes mellitus with clinically proved peripheral neuropathy. And control group (B) 40 patients with asymptomatic type 2 diabetes mellitus. They will be selected from South valley university hospitals. Group A will receive low intensity extracorporeal shock wave therapy for two per week for four weeks. Group B will receive shame low intensity extracorporeal shock wave therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitoring Effect Of Shock Wave On Microcirculation Changes In Type2 Diabetes Mellitus (Experimental): Energy intensity of (0.09 mJ/mm2) for 12 treatment sessions, two per week, for six weeks
  Interventions: Device: Low intensity extracorporeal shock wave
- Effect Of Shock Wave On Microcirculation Changes In Type2 Diabetes Mellitus (Experimental): low intensity extracorporeal shock wave with the following parameters: - 3000 SWs (energy intensity of (0.09 mJ/mm2).
  Interventions: Device: Low intensity extracorporeal shock wave

INTERVENTIONS:
Device: Low intensity extracorporeal shock wave — Extracorporeal shock wave therapy generator: Wonjin beauty SW10 shock wave therapy system made in Korean.
  Other Names: Shock wave

SUMMARY:
The purpose of the study is to monitor the effect of low intensity extracorporeal shock wave therapy on impaired nitric oxide synthase and microcirculation changes in type 2 diabetes mellitus with peripheral neuropathy.

DETAILED DESCRIPTION:
Low-intensity extracorporeal shockwave therapy (Li-ESWT) improved peripheral nerve repair and regeneration. Li-ESWT exerts its biological effects by increasing neuro¬trophic factors, Schwann cell activation, and cellular signaling activation. Li-ESWT could be a novel treatment for nerve injury-induced diabetic neuropathy and other conditions related to nerve in¬jury.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be symptomatically stable with type 2 diabetes mellitus complicated with peripheral neuropathy.
* Optimized pharmacological treatment that will be remained unchanged throughout the study.

Exclusion Criteria:

* Implanted cardiac pacemakers.
* Patients with known skin allergies.
* Presence of skin inflammations.
* Peripheral vascular disease.
* Patients with unstable angina pectoris.
* Progressive ventricular dysrhythmia.
* Intermittent claudication.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
• Nitric oxide level and electrophysiological investigations of peripheral nerves and muscles was measured pre and post treatment. | six weeks
  1. Laboratory methods: Nitric oxide laboratories for measurement of nitric oxide level.3. Electrodiagnostic studies are sensitive, specific, and validated measures of the presence of polyneuropathy.
• Numerical Rating Pain Scale | six weeks
  • The Numerical Rating Scale (NRS) is designed for anyone over age 9. It is one of the most commonly used pain scales in health care. To use it, you just say the number that best matches the level of pain you are feeling; you can also place a mark on the scale itself. Zero means you have no pain, while 10 represents the most intense pain possible.

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Luxor, South Valley University, Egypt

REFERENCES:
- [Background] Ovayolu N, Akarsu E, Madenci E, Torun S, Ucan O, Yilmaz M. Clinical characteristics of patients with diabetic polyneuropathy: the role of clinical and electromyographic evaluation and the effect of the various types on the quality of life. Int J Clin Pract. 2008 Jul;62(7):1019-25. doi: 10.1111/j.1742-1241.2008.01730.x. Epub 2008 Apr 10. PMID 18410351
- [Background] Cvijanovic M, Ilin M, Slankamenac P, Horvat SB, Jovin Z. The sensitivity of electromyoneurography in the diagnosis of diabetic polyneuropathy. Med Pregl. 2011 Jan-Feb;64(1-2):11-4. doi: 10.2298/mpns1102011c. PMID 21545063